CLINICAL TRIAL: NCT06450795
Title: Effectiveness of High Intensity Electromagnetic Therapy and Pelvic Floor Exercises in Women With Urinary Incontinence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, mehtap kilicoz, PhD student, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-2981
Record Dates: First submitted 2024-06-05; First posted 2024-06-10 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Urinary Incontinence
Keywords: electromagnetic stimulation; urinary incontinence; pelvic floor muscle training
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High intensity functional electromagnetic stimulation (HIFEM) treatment group (Experimental): Participants in both groups will then receive PTKE treatment for 8 weeks, 3 days a week for 30-45 minutes, under the supervision of specialist physiotherapists. Additionally, Participants will also receive HIFEM treatment for 6 weeks, 2 days a week for 28 minutes. The evaluations will be repeated at the end of the treatment.
  Interventions: Behavioral: Participants in both groups will then receive PTKE treatment for 8 weeks, 3 days a week for 30-45 minutes, under the supervision of specialist physiotherapists.
- Pelvic floor muscle training group (Experimental): Participants in both groups will then receive PTKE treatment for 8 weeks, 3 days a week for 30-45 minutes, under the supervision of specialist physiotherapists.
  Interventions: Behavioral: Participants in both groups will then receive PTKE treatment for 8 weeks, 3 days a week for 30-45 minutes, under the supervision of specialist physiotherapists.

INTERVENTIONS:
Behavioral: Participants in both groups will then receive PTKE treatment for 8 weeks, 3 days a week for 30-45 minutes, under the supervision of specialist physiotherapists. — HIFEM treatment for 6 weeks, 2 days a week for 28 minutes. The evaluations will be repeated at the end of the treatment.
  Other Names: high intensity functional electromagnetic stimulation

SUMMARY:
The aim of this study is to evaluate the effect of pelvic floor exercises and high intensity electromagnetic therapy on pelvic floor muscle function, quality of life and urinary parameters in women with stress urinary incontinence. The individuals to be included in the study will be selected from women with stress urinary incontinence who receive follow-up from Medipol Acıbadem Hospital. Women who meet the inclusion criteria will be explained the details of the study by the responsible researcher and an informed consent form will be presented. The study is planned as two groups:

Group 1: Pelvic floor muscle training (PBST) group. Group 2: Pelvic floor muscle training and high intensity functional electromagnetic stimulation (HIFEM) treatment group.

Envelope opening method will be used for randomisation of the participants into two groups. They will be included in the first or second group according to the number in the envelope they choose.

Each participant will be given a baseline assessment. Participants in both groups will then receive PTKE treatment for 8 weeks, 3 days a week for 30-45 minutes, under the supervision of specialist physiotherapists. Participants in 2 groups will also receive HIFEM treatment for 6 weeks, 2 days a week for 28 minutes. The evaluations will be repeated at the end of the treatment.

Research Outcome Measures:

Demographic and Clinical Characteristics International Incontinence Consultation Questionnaire-Short Form Urogenital Distress Inventory (UDI-6) Quality of Life King Health Survey Muscle function Emg-Biofeedback

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as stress urinary incontinence by a physician,
* Between the ages of 20-65,
* Has not had recurrent vaginitis infection,
* Women with no active urinary tract infection or more than 3 urinary tract infections in the last 1 year will be included in the study.

Exclusion Criteria:

* History of cardiac implant or untreated cardiac arrhythmia,
* The presence of a metal implant,
* Vaginal and pelvic surgery within the last 6 months,
* Gave birth within the last 12 weeks and had a history of miscarriage within 6 weeks,
* A recent surgical procedure,
* Any concurrent UI treatment,
* With renal and hepatic insufficiency,
* Neurological or neuromuscular disease
* It will be excluded in case of any contraindication listed in the investigational device manual.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
International Incontinence Consultation Questionnaire-Short Form | 5 minute
  Urinary incontinence symptom severity and its effect on quality of life will be evaluated with the ICIQ-SF, the reliability and validity of the Turkish version of which was performed by Çetinel et al. The scale consists of a total of 6 items questioning the type, frequency and amount of urinary incontinence and the effects of incontinence on the individual's life. The scores that can be obtained from the scale vary between 0-21 and a higher score indicates an increase in the severity of incontinence.
Urogenital Distress Inventory (UDE-6) | 5 minute
  The UDI-6 consists of 6 questions and is graded with a 4-point Likert-type score. A minimum score of 0 is obtained from the UDE-6 and this means that 'the patient is not disturbed at all', while the maximum score of 18 means that 'the patient is extremely disturbed by the symptoms'. The scores are converted to a percentage and the score is determined. The higher the score, the greater the severity of the symptoms.
King's Health Questionnaire | 5 minute
  The reliability and validity of the Turkish version of the quality of life related to urinary symptoms will be evaluated with the KSA, which was studied by Kaya et al. The KSA consists of two parts and includes 32 items. The best score that can be obtained from the complaint severity scale is '0' and the worst score is '30', while the best score that can be obtained from the answers given to all KSA sub-section problems is '0' and the worst score is '100'.
EMG-Biofeedback | 5 minute
  Used to evaluate pelvic floor muscle activation

IPD SHARING:
Plan to Share IPD: No